CLINICAL TRIAL: NCT02729064
Title: Effect of Intranasal Insulin Administration on Glycaemia and Insulin Concentrations in Plasma and Cerebrospinal Fluid During Surgery
Brief Title: Intraoperative Nasal Insulin Effect on Plasma and CSF Insulin Concentration and Blood Glucose
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hiroaki Sato, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Hiroaki Sato, MD., PhD., Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 5381
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Ischemic Heart Disease; Aortic Aneurysm
Keywords: Intranasal Insulin; Insulin concentration; Blood glucose; Cerebro Spinal Fluid insulin; Intraoperative blood glucose; Cardiac Surgery; Thoracic Surgery
MeSH Terms: conditions — Myocardial Ischemia; Aortic Aneurysm | interventions — Insulin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intranasal 40 (Experimental): Patients will receive 40 IU of intranasal insulin (Humulin R) via a metered nasal dispenser
  Interventions: Drug: Humulin R
- Intranasal 80 (Experimental): Patients will receive 80 IU of intranasal insulin (Humulin R) via a metered nasal dispenser
  Interventions: Drug: Humulin R
- Placebo (Placebo Comparator): Patients will receive intranasal normal saline via a metered nasal dispenser
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Humulin R — Study subjects will receive intranasal insulin (Humulin R) via a metered nasal dispenser.
  Arms: Intranasal 40; Intranasal 80
Drug: Normal Saline — Study subjects will receive intranasal placebo (normal saline) via a metered nasal dispenser.
  Arms: Placebo

SUMMARY:
Intranasal insulin is reported to improves memory performance in patients suffering from cognitive impairment. The investigators have previously shown that intraoperative insulin administration preserves both short and long-term memory function after cardiac surgery. Applying intranasal insulin bypasses blood-brain barrier and cause elevation of insulin concentrations in the cerebrospinal fluid without major effects on peripheral insulin level. Patients undergoing major surgery are exposed to carbohydrate and insulin metabolism alteration. The goal of the study is to study the effect of intranasal insulin on blood glucose, plasma and cerebrospinal insulin concentration in patients undergoing cardiac surgery or endovascular thoracic aneurysm repair.

DETAILED DESCRIPTION:
Clinical trials have demonstrated that intranasal insulin improves both memory performance and metabolic integrity of the brain in patients suffering from Alzheimer's disease or cognitive impairment. A single dose of intranasal insulin acutely improved memory in memory-impaired older adults. Cognitive impairment in post-operative period is an increasing problem as more elderly patients undergo major surgery. The investigators have previously shown that intraoperative insulin administration while maintaining normoglycaemia preserves both short and long-term memory function after open heart surgery.

Applying insulin as a nasal spray bypasses blood-brain barrier and cause significant and sustained elevation of insulin concentrations in the cerebrospinal fluid (CSF) without major effects on peripheral insulin levels. The administration of 40 IU of intranasal insulin(INI) rapidly increases CSF insulin concentration within seven minutes, peaking after 30 minutes and remaining elevated for more than 80 minutes.

Presently it is not clear if CNS insulin plays a relevant role in controlling blood glucose in humans.

Patients undergoing major surgery are exposed to metabolic and endocrine alterations in carbohydrate, protein, and insulin metabolism, often summarized as the catabolic stress response. While the effect of intravenous insulin on glucose metabolism during surgery has been extensively studied the influence of intranasal insulin administration on intraoperative plasma insulin and blood glucose concentrations is unknown.

Goal and Objectives The goal of the present study is to study the effect of intranasal insulin on

* blood glucose and plasma insulin concentrations in patients undergoing elective cardiac surgery
* blood glucose, plasma insulin and cerebrospinal insulin concentration in patients undergoing elective endovascular thoracic aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

All patients (>18 years) undergoing elective open heart surgery requiring CPB or elective endovascular thoracic aortic aneurysm repair at the RVH.

Exclusion Criteria:

1. Planned use of drugs that effect plasma glucose concentration during the first four hours of surgery.
2. Patients with allergy to insulin
3. Patients with a base line blood glucose less than 3.9 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | During Surgery
  Arterial blood samples will be collected every 10 to 30 minutes during the surgery. Circulating concentrations of glucose will be measured.
Plasma Insulin | During Surgery
  Arterial blood samples will be collected every 10 to 30 minutes during the surgery. Plasma insulin will be measured.
Cerebrospinal Fluid Insulin | During Surgery
  Cerebrospinal Fluid will be taken every 10 to 30 minutes during the endovascular thoracic aneurysm repair surgery. Insuring concentration of Cerebrospinal fluid will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roque P, Nakadate Y, Sato H, Sato T, Wykes L, Kawakami A, Yokomichi H, Matsukawa T, Schricker T. Intranasal administration of 40 and 80 units of insulin does not cause hypoglycemia during cardiac surgery: a randomized controlled trial. Can J Anaesth. 2021 Jul;68(7):991-999. doi: 10.1007/s12630-021-01969-5. Epub 2021 Mar 15. PMID 33721199
- [Derived] Nakadate Y, Sato H, Roque P, Sato T, Matsukawa T, Wykes L, Kawakami A, Schricker T. Accuracy of blood glucose measurements using the NOVA StatStrip(R) glucometer during cardiac surgery: a prospective observational study. Can J Anaesth. 2019 Aug;66(8):943-952. doi: 10.1007/s12630-019-01350-7. Epub 2019 Mar 20. PMID 30895515